CLINICAL TRIAL: NCT04170530
Title: Neoadjuvant mFOLFOXIRI Chemotherapy Alone for Extramural Vascular Invasion(EMVI) Positive Rectal Cancer: A Phase II, Single-arm, Prospective Clinical Study
Brief Title: Neoadjuvant mFOLFOXIRI Chemotherapy Alone for Extramural Vascular Invasion Positive Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hanju Hua, Associate chief physician, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRICHEMO
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Extramural Vascular Invasion; Neoadjuvant; chemotherapy; mFOLFOXIRI
MeSH Terms: interventions — Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- mFOLFOXIRI (Experimental): patients received FOLFOXIRI alone for 6 cycles before surgery.
  Interventions: Drug: mFOLFOXIRI

INTERVENTIONS:
Drug: mFOLFOXIRI — irinotecan* 135 mg/m² + oxaliplatin 68 mg/m² + leucovorin 400 mg/m² + 5-FU 2400 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle
  Other Names: 5-FU; Oxaliplatin; Irinotecan

SUMMARY:
Extramural Vascular Invasion Positive(EMVI+) is a high risk of distant metastasis for locally advanced rectal cancer(LARC) after resection. The study is to evaluate the efficacy and safety of mFOLFOXIRI as neoadjuvant chemotherapy alone for EMVI+ LARC.

DETAILED DESCRIPTION:
It is an investigator-initiated, single institution, prospective, single-arm clinical study to evaluate the efficacy and safety of FOLFOXIRI as neoadjuvant chemotherapy alone for EMVI+ LARC.Patients of LARC with EMVI+ evaluated by pelvic magnetic resonance imaging (MRI) were enrolled in this trial. All EMVI+ LARC will receive the study regimen every 2 weeks for 6 cycles. MRI will be performed after 3 cycles of chemotherapy to assess clinical response.MRI was performed to assess clinical response after chemotherapy. Patients with mesorectal fascia-positive or ycT4a/b after re-evaluation would receive radiation before surgery, whereas responders would have immediate total mesorectal excision (TME).If the tumor response is good enough(partial response or complete response), the patient will receive another 3 cycles of FOLFOXIRI then surgery. On the contrary, if the tumor shows poor response(stable disease or progressive disease) or with mesorectal fascia-positive or ycT4a/b after re-evaluation, radiotherapy will be performed combined with capecitabine before operation. All patients will receive 6 cycles of mFOLFOX6 or 4 cycles XELOX as adjuvant chemotherapy after TME.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 to 75 years at diagnosis;
2. ECOG status 0 or 1;
3. Signed informed consent; able to comply with study and/or follow- up procedures;
4. Diagnosis of rectal adenocarcinoma;
5. Distal border of the tumor must be located < 12 cm from the anal verge;
6. MRI examination diagnosed EMVI-positive;
7. Tumor amenable to curative resection;
8. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment: (1) Neutrophilic granulocytes ≥ 3.0 x10^9/L, Platelet count ≥ 75 x 10^9/L, Hemoglobin (Hb) ≥ 90g/L; (2) bilirubin ≤1.5 x the upper limit of normal (ULN),Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) ≤ 2.5 x ULN; (3) Serum creatinine ≤ 1.5 x ULN.
9. No renal disease that would preclude study treatment or follow-up

Exclusion Criteria:

1. Hypersensitivity to fluorouracil, oxaliplatin or irinotecan;
2. Patient had received pelvic radiotherapy;
3. Patient had received systemic chemotherapy;
4. History of invasive colon or rectal malignancy, regardless of disease-free interval;
5. Had metastatic disease;
6. Patient had second malignant disease within 5 years;
7. Uncontrolled co-morbid illnesses or other concurrent disease;
8. Patients refused to signed informed consent.
9. Pregnant and Nursing women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
MFS | Three years
  metastasis free survival

SECONDARY OUTCOMES:
Tumor downstaging rate | 2 years
  the proportion of tumor downstaging to ypT0-2N0M0
pCR | 2 years
  Pathologic complete response rate
R0 rate | 2 years
  R0 resection rate
locoregional recurrence | 3 years
  The rate of local recurrence
DFS | 3 years
  disease-free survival
OS | 5 years
  overall survival.
Reported Adverse events | 2 years
  The incidence of >=3 grade adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No